CLINICAL TRIAL: NCT06481527
Title: The Seen and Be Heard Study: Identifying the Barriers and Facilitators to Ensuring Equitable Cancer Care for Children With and Without a Learning Disability and/or Autism Spectrum Condition.
Brief Title: Seen and Be Heard: Ensuring Fair Cancer Care for All Children
Status: Not yet recruiting | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 22CB16
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Oncology; Haematological Malignancy
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children and young people: Children and young people aged 5-15 with or without learning disabilities or autism that are receiving cancer care.
- Parents: Parents of eligible children and young people aged 5-15 with or without learning disabilities or autism that are receiving cancer care.
- Healthcare Staff: Healthcare staff that provide cancer care services to children and young people.

SUMMARY:
Introduction:

Research has routinely been conducted into the experiences and well-being of children and young people with cancer and their families. However, there is little research that directly involves those with learning disabilities (LD) and or who are autistic. This is despite some cancers being more far more prevalent in some syndromes associated with learning disabilities, for example Downs Syndrome. More generally paediatric hospital care, recent research has highlighted inequity for children with LD, compared with children and young people without LD. Staff often feel less capable and confident to deliver care to those with learning disabilities, as well as having less capacity. Still less is known about cancer care for autistic children and young people, for example relating to symptom management. We aim to explore how inequity might present in cancer care for children and young people aged 5-15 years with and without LD and or who are autistic to see what inequities exist, for whom, why and in what circumstances.

Methods and analysis:

A transformative mixed methods design will be used, comprising an individual staff and organisational level survey, retrospective case note review, ethnographic observations of clinical care, family and staff interviews, and participatory workshops. The ethnographer will follow and observe individual children and their families. A 'toolbox' of creative participatory methods will be employed, including providing a co-designed research data collection journal to support elicitation of the child's perspective.

Ethics and Dissemination: The study will run from September 2024 to January 2026. Health Research Authority approval is granted (REC Reference no. 24/LO/0410 | IRAS Project ID: 335623) for work package 2 and 3 involving the ethnography, with interviews and workshops.

ELIGIBILITY:
Work package 1

A) National staff survey

Inclusion criteria:

* Healthcare professionals involved in cancer care delivery
* UK based

Exclusion criteria:

Outside stated of location

B) Organisational survey

Inclusion criteria:

- Clinical service leads

C) Anonymised retrospective electronic case note review

Inclusion criteria:

Children and Young aged 0-16 with Cancer diagnosis between April 2017 - present, within one large children's hospital site.

Work Package 2 - Ethnography study (including interviews)

Inclusion criteria

* Children and Young people receiving cancer care, with/without learning disability and or who are autistic at hospital research site
* Ages 5-15

Exclusion criteria

* Within palliative care at the time of recruitment
* Subject to child safeguarding proceedings
* Outside of stated age range
* Children who have not been disclosed their cancer diagnosis and where their family would prefer to maintain a complete non-disclosure approach

Parents:

Inclusion

* Of children receiving cancer care in hospital research site
* If included for interview only, child's age may be aged 0-16
* Conversational English

Exclusion - Has mental health difficulties that would impair ability to participate effectively or create an unmanageable risk e.g. psychosis

Healthcare professionals:

Inclusion

- Service providers of cancer care at hospital research site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The aim of this study is to recruit approximately up to 50 participants across the different groups within the ethnography work package with approximately equal healthcare professionals to parents / children and young people. Many participants will be involved only in interviews. For every child without LD/ASC, two children with LD/ASC will be recruited. Healthcare professionals that provide cancer care will make up approximately half of this sample and it will be ensured that they do not outnumber family participants. It is estimated up to 12-16 (6-8 with learning disability and or who are autistic and 4-6 without LD or autism) participants in the ethnography will be required, with a further 10 in-depth parent interviews. Staff interviews will be conducted with up to 25 staff members. This number will allow breadth of exploration while remaining feasible for this work package.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-02 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional Staff Survey | 6 months
  Purpose designed survey to provide staff perspectives around capacity, capability and confidence in delivering cancer care to children and young people with and without learning disabilities and or who are autistic.
Length of hospital stay | 2017-2023
  Relevant to retrospective electronic case note review
Mortality | 2017-2023
  Relevant to retrospective electronic case note review
Symptom management profiles: e.g. pain, constipation, nausea and vomiting | 2017-2023
  Relevant to retrospective electronic case note review
Cross-sectional Organisational Survey | 6 months
  Purpose designed survey to explore organisational level policies, training and implementation of interventions including making reasonable adjustments.

REFERENCES:
- [Derived] Oulton K, Wray J, Foo-Caballero M, Flynn S, Harniess P, Rao A, Gibson F. The seen and be heard study: A national mixed methods study to identify the barriers and facilitators to ensuring equitable cancer care for children with and without learning disabilities and/or who are autistic - Protocol Paper. PLoS One. 2025 Nov 19;20(11):e0333020. doi: 10.1371/journal.pone.0333020. eCollection 2025. PMID 41259352